CLINICAL TRIAL: NCT03110237
Title: A Multidimensional Inpatient Balance Training Class to Improve Functional Outcomes in Rehabilitation Inpatients With ABI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Marian Cayer, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H16-02866
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Brain Injuries, Traumatic; Cerebrovascular Trauma; Acute Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Cerebrovascular Trauma; Brain Injuries | interventions — Artifacts

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Balance Training (BT) class (Active Comparator): Group based circuit training class, 30 minute session, twice a week for three weeks
  Interventions: Other: Control Balance Training (BT) class
- Fallproof Balance Training (BT) class (Experimental): Group based balance training class based on the FallProof(TM) approach, 30 minute session , twice a week for three weeks
  Interventions: Other: Fallproof Balance Training (BT) class

INTERVENTIONS:
Other: Control Balance Training (BT) class — Circuit training class with 11 stations, including: step-ups, ball kicking, balance beam, sit to stand, walk and carry, tandem walking, walking over a mat, walking up a ramp, walking at different speeds, speed walk, dual task walking.
  Arms: Control Balance Training (BT) class
Other: Fallproof Balance Training (BT) class — There are four categories of exercises in this approach including: center of gravity control training (e.g. multi-directional weight shifts in standing, standing with altered base of support), multisensory training (e.g. standing on compliant surfaces, eyes open/closed), postural strategy training (e.g. resisted perturbation to facilitate ankle, hip or step strategy), and gait pattern variation training (e.g. walking with altered base of support , walking over and around obstacles). Each training category will be allocated 5 minutes with two exercises in each category. An additional 5 minutes will be allotted for games to challenge balance (balloon volleyball, pass the potato, circle soccer).There will be opportunity for group discussion and observational learning.
  Arms: Fallproof Balance Training (BT) class

SUMMARY:
Many survivors of acquired brain injury (ABI) suffer from decreased balance and increased risks of falls. Previous studies indicate that balance training improves balance, reduces falls, and increases walking speed and balance confidence. The purpose of this study is to determine if a multidimensional balance training based on the FallProof(TM) approach achieves better improvements in balance and walking performance than the current practice . Participants will be assigned to: 1)a task-oriented circuit training balance class (current practice), or 2) balance training class based on the FallProof(TM) approach. Standardized tests will determine if participating in balance training helps improve balance, walking speed and balance confidence.

DETAILED DESCRIPTION:
The purpose of this pilot research study is to determine if a balance training (BT) class based on the FallProof(TM) approach achieves better balance and mobility outcomes than the current practice. The FallProof's approach focuses on multiple components of balance impairment including multisensory, postural strategy and centre of gravity control training. Current practice is a task-oriented circuit training balance class.

ABI survivors may have muscle weakness, decreased coordination and sensory loss, which contribute to reduced balance, difficulty with functional mobility and activities of daily living. Balance control provides the foundation for a person's ability to stand, walk and function independently. Previous studies indicate that balance training (BT) improves balance, reduces falls, increases walking speed and balance self-efficacy for ABI patients .The Ottawa Panel Evidence-Based Clinical Practice Guidelines for ABI Rehabilitation supported the use of BT based on the research evidence. Interventions such as task-oriented training, multisensory training, trunk control training and perceptual exercises demonstrate positive effect on balance and mobility outcomes. To our knowledge, there are few studies that have examined a multidimensional approach to BT.

A systematic review concluded that exercises performed for 20-60 minutes, 3-4 times a week for 6-12 weeks can improve balance in ABI patients. However, Treacy et al demonstrated that inpatient BT for just 2 weeks can improve balance compared to a control group who received traditional exercise interventions.

At GF Strong Rehabilitation Center (GFS), the usual care provided to the ambulatory ABI patients consists of individualized one to one physiotherapy treatment, as well as a high level BT class. Currently, this BT class is a circuit training class that focuses on task-oriented gait exercises. FallProof balance training is a group- based approach that includes multisensory, postural strategy, centre of gravity control and gait pattern training. It was originally developed for older adults with impaired balance; but there is no research on the effectiveness of this approach for ABI patients. The FallProof approach has been introduced to the low level and intermediate level BT class at GFS, for ABI patients with sever and moderate balance impairments. These classes received positive feedback from patients and therapists. Patients reported improved functional mobility and confidence after attending the class. However, there was no functional outcome measurements collected to compare the effectiveness of the previous class and the new FallProof class. We plan to modify the current circuit training high level balance class with the FallProof approach in the spring of 2017. Before introducing the FallProof class, we would like to collect outcome measures with the current BT class for three months, and then collect collect data with the new class for comparison. We would like to determine if a multidimensional group based BT treatment approach is more effective at improving functional outcomes compared to the current practice.

ELIGIBILITY:
Inclusion Criteria:

1. inpatients admitted to GFS with a diagnosis of ABI;
2. medical stability
3. has the cognitive ability to understand and follow instructions and participate in a class setting
4. a Berg Balance Score of ≥52;
5. able to walk independently with or without a mobility aid.

Exclusion Criteria:

1) unable to attend class in a group setting and/or unable to follow instructions.

Ages: 16 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-04-10 (Estimated); Primary Completion 2017-11-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Community Balance and Mobility Scale (CB & M) | after attending balance class for 3 weeks
  A performance measure composed of 13 challenging tasks. Item scores range from 0 to 5 and reflect progressive task difficulty. All tasks performed without ambulation aides.

SECONDARY OUTCOMES:
Timed Up and Go Test (TUG) | after attending balance class for 3 weeks
  Timing how long it takes for patient to rise from a chair, walks 3 meters at a comfortable and safe pace, turns, walks back to the chair and sits down.
4 meters Gait Speed Test (GST) | after attending balance class for 3 weeks
  Measure time (in seconds) that it takes the patient to walk 4 meters. The patient should be at their usual speed during the entire 4 meter timed area. Use a 6 meter path, with the central 4 meters as the timed area. Patient may use any walking aid.
Falls Efficacy Scale (FES) | after attending balance class for 3 weeks
  A 10-item questionnaire for patients to rate their confidence in their ability to perform 10 daily tasks without falling as an indicator of how one's fear of falling impacts physical performance. Each item is rated from 1 ("very confident") to 10 ("not confident at all").

CONTACTS AND LOCATIONS:
Overall Officials: Marian Cayer, BSc, Principal Investigator — Vancouver Coastal Health
Locations (1):
- GF Strong Rehabilitation Center, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pollock A, Baer G, Campbell P, Choo PL, Forster A, Morris J, Pomeroy VM, Langhorne P. Physical rehabilitation approaches for the recovery of function and mobility following stroke. Cochrane Database Syst Rev. 2014 Apr 22;2014(4):CD001920. doi: 10.1002/14651858.CD001920.pub3. PMID 24756870
- [Background] Winter D. A.B.C.(Anatomy, Biomechanics and Control) of Balance During Standing and Walking. Waterloo: Waterloo Biomechanics; 1995.
- [Background] Annabel McDermott, OT; Nicol Korner-Bitensky, PhD OT; Norine Foley, BASc; Mark Speechley, PhD; Nancy M. Salbach, PhD, PT; Maxim Ben Yakov, BSc. PT; Robert Teasell, MD. (2012). Balance Training. Retrieved from http://www.strokengine.ca/intervention/balance-training/
- [Background] Lubetzky-Vilnai A, Kartin D. The effect of balance training on balance performance in individuals poststroke: a systematic review. J Neurol Phys Ther. 2010 Sep;34(3):127-37. doi: 10.1097/NPT.0b013e3181ef764d. PMID 20716987
- [Background] An M, Shaughnessy M. The effects of exercise-based rehabilitation on balance and gait for stroke patients: a systematic review. J Neurosci Nurs. 2011 Dec;43(6):298-307. doi: 10.1097/JNN.0b013e318234ea24. PMID 22089406
- [Background] Ottawa Panel; Khadilkar A, Phillips K, Jean N, Lamothe C, Milne S, Sarnecka J. Ottawa panel evidence-based clinical practice guidelines for post-stroke rehabilitation. Top Stroke Rehabil. 2006 Spring;13(2):1-269. doi: 10.1310/3TKX-7XEC-2DTG-XQKH. PMID 16939981
- [Background] Lindsay MP, Gubitz G, Bayley M, Hill MD, Davies-Schinkel C, Singh S, and Phillips S. Canadian Best Practice Recommendations for Stroke Care (Update 2010). On behalf of the Canadian Stroke Strategy Best Practices and Standards Writing Group. 2010; Ottawa, Ontario Canada: Canadian Stroke Network.
- [Background] Richards CL, Malouin F, Wood-Dauphinee S, Williams JI, Bouchard JP, Brunet D. Task-specific physical therapy for optimization of gait recovery in acute stroke patients. Arch Phys Med Rehabil. 1993 Jun;74(6):612-20. doi: 10.1016/0003-9993(93)90159-8. PMID 8503751
- [Background] McClellan R, Ada L. A six-week, resource-efficient mobility program after discharge from rehabilitation improves standing in people affected by stroke: placebo-controlled, randomised trial. Aust J Physiother. 2004;50(3):163-7. doi: 10.1016/s0004-9514(14)60154-9. PMID 15482247
- [Background] Yelnik AP, Le Breton F, Colle FM, Bonan IV, Hugeron C, Egal V, Lebomin E, Regnaux JP, Perennou D, Vicaut E. Rehabilitation of balance after stroke with multisensorial training: a single-blind randomized controlled study. Neurorehabil Neural Repair. 2008 Sep-Oct;22(5):468-76. doi: 10.1177/1545968308315996. PMID 18780882
- [Background] Alptekin N, Gok H, Geler-Kulcu D, Dincer G. Efficacy of treatment with a kinaesthetic ability training device on balance and mobility after stroke: a randomized controlled study. Clin Rehabil. 2008 Oct-Nov;22(10-11):922-30. doi: 10.1177/0269215508090673. PMID 18955424
- [Background] Karthikbabu S, Nayak A, Vijayakumar K, Misri Z, Suresh B, Ganesan S, Joshua AM. Comparison of physio ball and plinth trunk exercises regimens on trunk control and functional balance in patients with acute stroke: a pilot randomized controlled trial. Clin Rehabil. 2011 Aug;25(8):709-19. doi: 10.1177/0269215510397393. Epub 2011 Apr 19. PMID 21504955
- [Background] Sackley CM, Lincoln NB. Single blind randomized controlled trial of visual feedback after stroke: effects on stance symmetry and function. Disabil Rehabil. 1997 Dec;19(12):536-46. doi: 10.3109/09638289709166047. PMID 9442992
- [Background] Morioka S, Yagi F. Effects of perceptual learning exercises on standing balance using a hardness discrimination task in hemiplegic patients following stroke: a randomized controlled pilot trial. Clin Rehabil. 2003 Sep;17(6):600-7. doi: 10.1191/0269215503cr654oa. PMID 12971704
- [Background] Bonan IV, Yelnik AP, Colle FM, Michaud C, Normand E, Panigot B, Roth P, Guichard JP, Vicaut E. Reliance on visual information after stroke. Part II: Effectiveness of a balance rehabilitation program with visual cue deprivation after stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2004 Feb;85(2):274-8. doi: 10.1016/j.apmr.2003.06.016. PMID 14966713
- [Background] Treacy D, Schurr K, Lloyd B, Sherrington C. Additional standing balance circuit classes during inpatient rehabilitation improved balance outcomes: an assessor-blinded randomised controlled trial. Age Ageing. 2015 Jul;44(4):580-6. doi: 10.1093/ageing/afv019. Epub 2015 Mar 10. PMID 25758408
- [Background] Rose DJ. Reducing the risk of falls among older adults: the Fallproof Balance and Mobility Program. Curr Sports Med Rep. 2011 May-Jun;10(3):151-6. doi: 10.1249/JSR.0b013e31821b1984. PMID 21623303
- [Background] Ng SS, Hui-Chan CW. The timed up & go test: its reliability and association with lower-limb impairments and locomotor capacities in people with chronic stroke. Arch Phys Med Rehabil. 2005 Aug;86(8):1641-7. doi: 10.1016/j.apmr.2005.01.011. PMID 16084820
- [Background] van Hedel HJ, Wirz M, Dietz V. Assessing walking ability in subjects with spinal cord injury: validity and reliability of 3 walking tests. Arch Phys Med Rehabil. 2005 Feb;86(2):190-6. doi: 10.1016/j.apmr.2004.02.010. PMID 15706542
- [Background] Howe JA, Inness EL, Venturini A, Williams JI, Verrier MC. The Community Balance and Mobility Scale--a balance measure for individuals with traumatic brain injury. Clin Rehabil. 2006 Oct;20(10):885-95. doi: 10.1177/0269215506072183. PMID 17008340
- [Background] van Hedel HJ, Wirz M, Dietz V. Standardized assessment of walking capacity after spinal cord injury: the European network approach. Neurol Res. 2008 Feb;30(1):61-73. doi: 10.1179/016164107X230775. PMID 17767814
- [Background] Scivoletto G, Tamburella F, Laurenza L, Foti C, Ditunno JF, Molinari M. Validity and reliability of the 10-m walk test and the 6-min walk test in spinal cord injury patients. Spinal Cord. 2011 Jun;49(6):736-40. doi: 10.1038/sc.2010.180. Epub 2011 Jan 11. PMID 21221120
- [Background] Tyson S, Connell L. The psychometric properties and clinical utility of measures of walking and mobility in neurological conditions: a systematic review. Clin Rehabil. 2009 Nov;23(11):1018-33. doi: 10.1177/0269215509339004. Epub 2009 Sep 28. PMID 19786420
- [Background] Hellstrom K, Lindmark B. Fear of falling in patients with stroke: a reliability study. Clin Rehabil. 1999 Dec;13(6):509-17. doi: 10.1191/026921599677784567. PMID 10588538
- [Background] Medley A, Thompson M, French J. Predicting the probability of falls in community dwelling persons with brain injury: a pilot study. Brain Inj. 2006 Dec;20(13-14):1403-8. doi: 10.1080/02699050601082057. PMID 17378232
- [Background] Wirz M, Muller R, Bastiaenen C. Falls in persons with spinal cord injury: validity and reliability of the Berg Balance Scale. Neurorehabil Neural Repair. 2010 Jan;24(1):70-7. doi: 10.1177/1545968309341059. Epub 2009 Aug 12. PMID 19675123